CLINICAL TRIAL: NCT07131839
Title: Effects of Central Sensitization Presence on the Results of Shoulder Adhesive Capsulitis Treatment With Physical Therapy Agents and Exercise
Brief Title: Central Sensitization Presence on the Results of Shoulder Adhesive Capsulitis
Acronym: FrozenShoulder
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hüma Bölük Şenlikci, Associate Prof, Ankara City Hospital Bilkent
Other Study IDs: KA 21/47; AnkaraCHBilkent (Other: Başkent University Medical School Hospital)
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Adhesive Capsulitis of the Shoulder
Keywords: Adhesive Capsulitis; chronic pain
MeSH Terms: conditions — Bursitis; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Adhesive shoulder patients with central sensitization
- Group 2: Adhesive capsulitis patients without central sensitization

SUMMARY:
Patients with adhesive capulitis longlasting more than 3 months were participated in the study. they were divided into two groups whether they have central sensitizaiton or not. Conventional physical therapy responses were measured and compared between two groups.

DETAILED DESCRIPTION:
Adhesive capsulitis is a well known musculoskeletal syndrome that effects daily living activities and patiemts suffer from chronic shoulder pain. Central sensitization has been defined in patients with chronic pain due to amplified neuronal connections and signals in the central nervous system. Previously, it was shown that refractory long lasting musculoskeletal disorders may show challenging treatment process and decreased outcome due to central sensitization. However to the best of our knowledge there was not any study that evaluates the treatment response of presence of central sensitization in adhesive capsulitis patients. Total of 32 adhesive capsulitis patients were particapted in the study. Sixteen patients with adhesive capsulitis with (Group 1) and without central sensitization (Group 2) were received conventional physical therapy and exercise. Treatment response were evaluated with Visual Analog Scale (VAS), Shoulder pain and disability index (SPADI) Tampa Kinesiophobia Scale (TKS) and Pain Catastrophizing Scale (PCS). Additionally shoulder range of motion was measured at baseline (T0), after treatment (T1) and at 2nd week after completion of conventional rehabilitation program (T2).

ELIGIBILITY:
Inclusion Criteria:

1)patients with adhesive capsulitis between 18-80 years old 2) symptoms ongoing more than 3 months 3) willing to participated in the study

Exclusion Criteria:

1) patients with cervical radiculopathy 2) Patients with predisposing factors to adhesive capsulitis, such as diabetes mellitus, thyroid disease, coronary artery disease, lung pathologies or tuberculosis 3) any defined central sensitization syndrome such as fibromiyalgia before 4) presence of rheumatologic diseases 5) pregnancy 6) patients underwent bypass surgery or who have cardiac pacemaker 7) patients with septic arthritis or sepsis 8) malignancy 9) patients that underwent surgery through the shoulder region or had injection through the shoulder joint in the last 3 months.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adhesive capsulitis patients aged between 18-80 years, and symptoms ongoing more than 3 months were participated in the study
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | at baseline (T0), after treatment (T1) and at 2nd week after completion of conventional rehabilitation program (T2)
  A 10 cm VAS, with known validity and reliability, was used as a self-reported measure for the severity of joint pain.
Shoulder Pain Disability Index (SPADI) | at baseline (T0), after treatment (T1) and at 2nd week after completion of conventional rehabilitation program (T2)
  This questionnaire was developed to assess shoulder joint pain and disability. The SPADI has two sections; first section contains 5 questions to evaluate pain, whereas second item contains 8 questions to evaluate disability. Scores vary 0-130 and higher scores indicates high disability rates and pain
Measurement of Shoulder range of motion | at baseline (T0), after treatment (T1) and at 2nd week after completion of conventional rehabilitation program (T2)
  The same physician performed the measurement for the joint ranges in each plane of the joint with a goniometer. The goniometer's pivot point was positioned on the lateral projection of the shoulder joint while subjects in supine position. The fixed arm aligned parallel to the axillary lateral midline , while the movable arm tracked the humerus' lateral midline movement towards the axilla. The joint was passively forced to the end of the direction of range and measured twice and the average was taken

SECONDARY OUTCOMES:
Tampa Kinesiophobia Scale (TKS) | at baseline (T0), after treatment (T1) and at 2nd week after completion of conventional rehabilitation program (T2)
  It was used to measure pain and the resulting fear and avoidance of moving the painful body part. TKS contains 17 questions assess parameters of injury/re-injury and fear or avoidance in work-related activities. Scores vary 17-68 and higher scores indicates higher kinseiophobia levels
Pain Catastrophizing Scale (PCS) | at baseline (T0), after treatment (T1) and at 2nd week after completion of conventional rehabilitation program (T2).
  PCS was created to evaluate the perception of catastrophizing caused by pain. It provide an objective assessment of the cognitive status related to pain. It consists of a self-administered 13-question and Likert scale (0, means never; 4, means always) is used in scoring. Total score is between 0-52 and with higher scores, perception of catastrophizing increases
Beck Depression Inventory (BDI) | at baseline (T0), after treatment (T1) and at 2nd week after completion of conventional rehabilitation program (T2)
  Beck Depression Inventory (BDI) is used to evaluate the characteristics of depression and anxiety. BDI consists of 21 questions, higher scores imply increased depression symptom severity

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing is going to be considered after submitted to a journal

REFERENCES:
- [Background] Bilika P, Nijs J, Fandridis E, Dimitriadis Z, Strimpakos N, Kapreli E. In the Shoulder or in the Brain? Behavioral, Psychosocial and Cognitive Characteristics of Unilateral Chronic Shoulder Pain with Symptoms of Central Sensitization. Healthcare (Basel). 2022 Aug 30;10(9):1658. doi: 10.3390/healthcare10091658. PMID 36141270
- [Background] Brindisino F, Girardi G, Crestani M, Fiore A, Giovannico G, Garzonio F, Venturin D, Struyf F. Effectiveness of electrophysical agents in subjects with frozen shoulder: a systematic review and meta-analysis. Disabil Rehabil. 2024 Aug;46(16):3513-3534. doi: 10.1080/09638288.2023.2251880. Epub 2023 Sep 5. PMID 37667875
- [Background] James-Belin E, Lasbleiz S, Haddad A, Morchoisne O, Ostertag A, Yelnik A, Laredo JD, Bardin T, Orcel P, Richette P, Beaudreuil J. Shoulder adhesive capsulitis: diagnostic value of active and passive range of motion with volume of gleno-humeral capsule as a reference. Eur J Phys Rehabil Med. 2020 Aug;56(4):438-443. doi: 10.23736/S1973-9087.19.05890-8. Epub 2019 Nov 18. PMID 31742369